CLINICAL TRIAL: NCT00418041
Title: Chronic Heart Failure Analysis and Registry in the Tohoku District 2 (CHART-2 Study)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hiroaki Shimokawa, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Hiroaki Shimokawa, MD, PhD, Department of Cardiovascular Medicine, Tohoku University
Organization: Tohoku University (Other)
Other Study IDs: 2006-115
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Heart Failure; Coronary Disease; Heart Valve Diseases; Cardiomyopathies; Left Ventricular Hypertrophy
MeSH Terms: conditions — Heart Failure; Coronary Disease; Heart Valve Diseases; Cardiomyopathies; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic Heart Failure Analysis and Registry in the Tohoku District 2 (CHART-2 Study) is a large, prospective, hospital-based cohort study to investigate the following:

* Characteristics of patients with chronic heart failure and prognostic risks of these patients.
* Characteristics of patients with high risk for heart failure and critical factors which predict the development of symptomatic heart failure in these patients.
* The incidence and prognostic impact of metabolic syndrome in patients with chronic heart failure.
* The association between metabolic syndrome and the development of symptomatic heart failure.

DETAILED DESCRIPTION:
The CHART-2 Study is a multicenter prospective observational cohort study identifying the characteristics, mortality and prognostic risks of patients with overt HF and patients without HF but who are at high risk for disease progression of cardiovascular diseases (CVD).

The purposes of the study are as follows:

1. to elucidate characteristics of patients with overt HF and the associated prognostic risks
2. to elucidate characteristics of patients at risk for HF and the factors associated with CVD progression
3. to elucidate factors associated with the development of AHFS
4. to elucidate prevalence and prognostic impact of metabolic syndrome (MetS) in patients with overt HF
5. to elucidate the association between MetS and the development of AHFS
6. to elucidate the prevalence and prognostic impact of malignancy in patients with CVD
7. to elucidate the prevalence of patients needing home nursing care and the characteristics of bedridden patients with CVD.

ELIGIBILITY:
Inclusion Criteria:

* Structural heart disease but without signs or symptoms of heart failure.
* Structural heart disease with prior or current symptoms of heart failure.
* Refractory heart failure requiring specialized interventions.
* Patients with prior cardiovascular surgery or percutaneous coronary intervention and those who need such interventions.

Exclusion Criteria:

* Patients with age<20 years old.
* Patients who refused to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in teaching hospitals
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2006-10; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
All-cause death | At the time of registration and at least once a year thereafter
Non-fatal acute myocardial infarction | At the time of registration and at least once a year thereafter
Non-fatal stroke | At the time of registration and at least once a year thereafter
Heart failure requiring admission | At the time of registration and at least once a year thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Shimokawa, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Tohoku University Graduate School of Medicine, Sendai, Japan

REFERENCES:
- [Derived] Ito T, Nochioka K, Noda T, Shiroto T, Yamanaka S, Yamamoto N, Sato H, Chiba T, Nakano M, Inoue T, Susukita K, Takahama H, Takahashi J, Miyata S, Shimokawa H, Yasuda S. New-onset anemia and its association with ventricular arrhythmias and sudden cardiac death in patients with heart failure with preserved ejection fraction. Int J Cardiol Heart Vasc. 2025 Sep 25;61:101812. doi: 10.1016/j.ijcha.2025.101812. eCollection 2025 Dec. PMID 41069488
- [Derived] Ito T, Noda T, Nochioka K, Shiroto T, Yamamoto N, Sato H, Hayashi H, Chiba T, Nakano M, Takahama H, Takahashi J, Miyata S, Shimokawa H, Yasuda S. Association of a mild or an important decline in left ventricular ejection fraction with ventricular tachyarrhythmias, sudden cardiac death, and all-cause death in heart failure with preserved ejection fraction: a report from the CHART-2 Study. Europace. 2025 Sep 1;27(9):euaf184. doi: 10.1093/europace/euaf184. PMID 40879292
- [Derived] Ito T, Noda T, Nochioka K, Shiroto T, Yamamoto N, Sato H, Chiba T, Hasebe Y, Nakano M, Takahama H, Takahashi J, Miyata S, Shimokawa H, Yasuda S. Clinical impact of atrial fibrillation progression in patients with heart failure with preserved ejection fraction: A report from the CHART-2 Study. Europace. 2024 Aug 30;26(9):euae218. doi: 10.1093/europace/euae218. PMID 39150084
- [Derived] Aoyanagi H, Nochioka K, Sakata Y, Miura M, Shiroto T, Abe R, Kasahara S, Sato M, Fujihashi T, Yamanaka S, Hayashi H, Sugimura K, Takahashi J, Miyata S, Shimokawa H; CHART-2 Investigators. Temporal changes in left ventricular ejection fraction and their prognostic impacts in patients with Stage B heart failure. Int J Cardiol. 2020 May 1;306:123-132. doi: 10.1016/j.ijcard.2020.02.040. Epub 2020 Feb 15. PMID 32113664
- [Derived] Takada T, Sakata Y, Nochioka K, Miura M, Abe R, Kasahara S, Sato M, Aoyanagi H, Fujihashi T, Yamanaka S, Suzuki K, Shiroto T, Sugimura K, Takahashi J, Miyata S, Shimokawa H; CHART-2 Investigators. Risk of de-novo heart failure and competing risk in asymptomatic patients with structural heart diseases. Int J Cardiol. 2020 May 15;307:87-93. doi: 10.1016/j.ijcard.2020.02.015. Epub 2020 Feb 6. PMID 32107021
- [Derived] Suzuki K, Oikawa T, Nochioka K, Miura M, Kasahara S, Sato M, Aoyanagi H, Shiroto T, Takahashi J, Miyata S, Sakata Y, Shimokawa H. Elevated Serum Non-HDL (High-Density Lipoprotein) Cholesterol and Triglyceride Levels as Residual Risks for Myocardial Infarction Recurrence Under Statin Treatment. Arterioscler Thromb Vasc Biol. 2019 May;39(5):934-944. doi: 10.1161/ATVBAHA.119.312336. PMID 30866657
- [Derived] Oikawa T, Sakata Y, Nochioka K, Miura M, Tsuji K, Onose T, Abe R, Kasahara S, Sato M, Shiroto T, Takahashi J, Miyata S, Shimokawa H; CHART-2 invesigators. Prognostic Impact of Statin Intensity in Heart Failure Patients With Ischemic Heart Disease: A Report From the CHART-2 (Chronic Heart Failure Registry and Analysis in the Tohoku District 2) Study. J Am Heart Assoc. 2018 Mar 14;7(6):e007524. doi: 10.1161/JAHA.117.007524. PMID 29540427
- [Derived] Ushigome R, Sakata Y, Nochioka K, Miyata S, Miura M, Tadaki S, Yamauchi T, Sato K, Onose T, Tsuji K, Abe R, Oikawa T, Kasahara S, Takahashi J, Shimokawa H; CHART-2 Investigators. Temporal trends in clinical characteristics, management and prognosis of patients with symptomatic heart failure in Japan -- report from the CHART Studies. Circ J. 2015;79(11):2396-407. doi: 10.1253/circj.CJ-15-0514. Epub 2015 Sep 10. PMID 26356834
- [Derived] Miura M, Sakata Y, Miyata S, Nochioka K, Takada T, Tadaki S, Takahashi J, Shiba N, Shimokawa H; CHART-2 Investigators. Usefulness of combined risk stratification with heart rate and systolic blood pressure in the management of chronic heart failure. A report from the CHART-2 study. Circ J. 2013;77(12):2954-62. doi: 10.1253/circj.cj-13-0725. Epub 2013 Oct 1. PMID 24088306